CLINICAL TRIAL: NCT02970331
Title: A Phase 2, Multicenter, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Pefcalcitol Ointment, 0.005%, Applied Topically Twice Daily (BID) for 8 Weeks in Adolescent Subjects 12 to < 17 Years of Age With Plaque Psoriasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA requested us to stop the study
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLS008-CO-PR-001
Record Dates: First submitted 2016-11-16; First posted 2016-11-22 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- pefcalcitol (Experimental): pefcalcitol 0.005% BID for 8 weeks
  Interventions: Drug: pefcalcitol ointment, 0.005%

INTERVENTIONS:
Drug: pefcalcitol ointment, 0.005% — pefcalcitol ointment, 0.005%

SUMMARY:
A multi-center, open-label study that will evaluate the safety/tolerability and pharmacodynamics as well as the pharmacokinetic profile (sub-population analysis), in 50 evaluable adolescents 12 to < 17 years of age.

ELIGIBILITY:
Inclusion Criteria:

* male or females 12 to < 17 years of age
* Have a confirmed diagnosis of plaque psoriasis
* Negative pregnancy test
* Group 1: Have plaque psoriasis with an IGA score of ≥ 2 (mild), with at least one lesion ) and up to 20% Body Surface Area (BSA) involvement not including psoriasis on the face and scalp
* Group 2: Have plaque psoriasis with a IGA score of ≥ 2 (mild), with plaque psoriasis involving at least 10% and up to 20% Body Surface Area (BSA) not including psoriasis on the face and scalp

Exclusion Criteria:

* known allergy or intolerance to the study drug or other vitamin D3 analogs or any of its components
* history of or active generalized guttate, pustular or erythrodermic exfoliative psoriasis
* history or presence of contact dermatitis induced by a topical medicine or other serious skin condition that is not well controlled
* Use topical treatments known to have beneficial effects on psoriasis
* Use phototherapy, oral corticosteroids, oral retinoid, oral immunosuppressive/immunomodulate drugs, cytostatics, cyclosporine or methotrexate within 30 days prior to the first dose of study drug
* Use any approved biologics for psoriasis within 30 days or 5 half-lives of the biologic before the first dose of study drug
* Are treated with medications known to worsen psoriasis
* Are taking an oral vitamin D
* Are taking medications that affect calcium metabolism;
* Subjects who have an average of three (3) QTcF measurements of > 450 milliseconds as shown on the ECG (Group 2 only);
* Have clinically significant abnormal calcium homeostasis parameters at Visit 1;
* Have clinically significant liver or renal dysfunction
* Have any other clinically significant laboratory abnormalities, co-morbidities or psychiatric conditions which that would place the subject at increased risk or would confound the primary or secondary objectives of the study;
* Use of any investigational drugs or biologics and/or participated in any clinical trial within the last 60 days before the day of the first dose of study drug or are taking part in a non-medication study which, that would interfere with study compliance or outcome assessments;
* Are pregnant or lactating females;
* Have a known history of congenital or acquired immunodeficiency.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in incidence and severity of application site adverse events | screening, weeks 0,2,4 and 8
Change in incidence and severity of all AEs and their relationship to study drug | screening, weeks 0,2,4 and 8
Changes from baseline (pre-dose, Day 1) in safety laboratory parameters | week 8
Changes from baseline (pre-dose, Day 1) in calcium homeostasis parameters (total serum calcium and albumin-corrected calcium levels, plasma parathyroid hormone (PTH), and serum alkaline phosphatase) | week 8
Determination of plasma concentrations of Pefcalcitol and its metabolites | Day 1 and Day 15

SECONDARY OUTCOMES:
Proportion of subjects with an IGA score of absence (0) or very mild (1) with a minimum of a 2-grade improvement from baseline | week 8
Proportion of subjects who achieved an mPASI 75 from baseline (Week 0) to Week 8, or who achieved an mPASI 50 and a 5-point improvement in the CDLQI from baseline | week 8
Proportion of subjects who achieved success in each of the three individual components of the mPASI (scaling, thickness and erythema) from baseline | week 8
Proportion of subjects who achieved a 5-point improvement in the CDLQI from baseline | week 8